CLINICAL TRIAL: NCT06196541
Title: Edema, Pain, Respiratory Functions, Physical Functions and Quality of Life in Individuals With Chronic Venous Insufficiency
Brief Title: Respiratory and Physical Functions in Individuals With Chronic Venous Insufficiency
Status: Active, not recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Assoc.Prof., Izmir Democracy University
Other Study IDs: Chronic venous insufficiency
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Chronic Venous Insufficiency
Keywords: edema; pain; venous insufficiency; quality of life; respiratory function tests; maximal respiratory pressures; exercise capacity
MeSH Terms: conditions — Edema; Pain; Venous Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Chronic Venous Insufficiency: Edema, pain, respiratory functions, physical functions and quality of life will be evaluated in individuals with chronic venous insufficiency.
- Asymptomatic Healthy Individuals: Edema, pain, respiratory functions, physical functions and quality of life will be evaluated in asymptomatic healthy individuals.

SUMMARY:
In the literature, it is still unclear whether individuals with chronic venous insufficiency are affected by edema, pain, respiratory muscle strength, respiratory functions, functional capacity, lower extremity strength and quality of life compared to asymptomatic healthy individuals and if there is a deterioration in these parameters, its level is still unclear. For this reason, in this study it was aimed to investigate edema, pain, respiratory muscle strength, respiratory function, functional capacity, lower extremity strength and quality of life in individuals with chronic venous insufficiency and asymptomatic healthy individuals and to compare these parameters between the two groups.

DETAILED DESCRIPTION:
Chronic Venous Insufficiency affects approximately 30% of the global population and its main symptoms are pain, edema, throbbing, feeling of heaviness in the extremities, itching, varicose veins and tissue changes. Pain in CVI is a chronic condition that negatively affects the quality of life due to physical function and limitation of movement. Limitation of ankle movement in CVI is one of the factors that increase edema and venous severity. Fibrotic tissue formations in the lower extremity cause limitation in ankle movements. In a study by De Moura et al. it was found that walking speed, muscle strength and functional capacity levels of patients with chronic venous insufficiency were limited compared to healthy individuals. Venous function is reflected from venous return, venous resistance and its effects on cardiac output. Venous filling time is a parameter of venous function and is shortened as a result of valve insufficiency, vessel wall dilatation and muscle pump dysfunction. The calf muscles compress the deep intramuscular veins, directing blood flow from the veins to the heart. However, muscle pump dysfunction is not limited to the calf muscle but also includes inspiratory muscle dysfunction. It is known that the diaphragm creates a suction effect in the inferior vena cava during inspiration and expiration, allowing more blood flow from the lower extremities to the heart. The respiratory cycle has been shown to affect venous return in healthy individuals by increasing deep inspiration and the flow rate of the femoral vein. Researches investigating pulmonary function in chronic venous insufficiency are very limited. For this reason, in this study it was aimed to investigate edema, pain, respiratory muscle strength, respiratory function, functional capacity, lower extremity strength and quality of life in individuals with chronic venous insufficiency and asymptomatic healthy individuals and to compare these parameters between the two groups.

ELIGIBILITY:
Inclusion criteria for individuals with chronic venous insufficiency:

* Being diagnosed with chronic venous insufficiency
* Being in one of the C1, C2, C3, C4, C5 stages according to the 'Clinical, Etiologic, Anatomic, Pathophysiologic' (CEAP) scale
* Volunteering to participate in the study
* 18 years of age or older

Exclusion criteria for individuals with chronic venous insufficiency:

* Presence of arterial disease,
* The presence of advanced cardiorespiratory diseases,
* Orthopaedic and neurological disorders affecting walking,
* Presence of acute ulcers (< 3 months) and diabetic ulcers,
* Being pregnant.
* History of deep vein thrombosis,
* Presence of active infection

Inclusion criteria for asymptomatic healthy individuals:

* 18 years of age and older
* Volunteering to participate in the study
* Individuals who can understand and answer questionnaires and measurements

Exclusion criteria for asymptomatic healthy individuals:

* Individuals with any physical or mental disability
* Individuals with any acute or chronic infection and/or health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer adult individuals diagnosed with chronic venous insufficiency by a Cardiovascular Specialist and healthy volunteer adult individuals without a diagnosis of chronic venous insufficiency will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2026-12-27 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | through study completion, an average of 1 year
  The MIP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.
Maximal expiratory pressure (MEP) | through study completion, an average of 1 year
  The MEP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.

SECONDARY OUTCOMES:
Pain Intensity measured with the Numerical Rating Scale. | through study completion, an average of 1 year
  Pain intensity will be measured with the Numerical Rating Scale. This scale expresses the severity of pain with integers from 0 (no pain) to 10 (the worst possible pain).
The distance of six-minute walk test | through study completion, an average of 1 year
  The six-minute walk test (6-MWT) will be performed according to the criteria of the American Thoracic Society for the evaluation of aerobic capacity.
Lower extremity strength | through study completion, an average of 1 year
  To determine lower extremity strength and functional mobility, the 30-second Sit-Up Test will be used in the chair.
Total quality of life score evaluated by Chronic Venous Disease Quality of Life Questionnaire | through study completion, an average of 1 year
  The score will be evaluated using Chronic Venous Disease Quality of Life Questionnaire. Each question is scored on a 5-item Likert scale. Higher scores indicate better quality of life.
Forced vital capacity (FVC) | through study completion, an average of 1 year
  Pulmonary function (Forced vital capacity (FVC) will be evaluated with a spirometer.
Forced expiratory volume in the first second (FEV1) | through study completion, an average of 1 year
  Pulmonary function (Forced expiratory volume in the first second (FEV1) will be evaluated with a spirometer.
FEV1 / FVC | through study completion, an average of 1 year
  Pulmonary function (FEV1 / FVC) will be evaluated with a spirometer.
Flow rate 25-75% of forced expiratory volume (FEF 25-75%) | through study completion, an average of 1 year
  Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated with a spirometer.
Peak flow rate (PEF) | through study completion, an average of 1 year
  Pulmonary function (Peak flow rate (PEF) will be evaluated with a spirometer.
edema | through study completion, an average of 1 year
  Edema in the lower extremity will be evaluated by measuring the circumference using a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Assoc. Dr., Study Director — Izmir Democracy University; ÖZLEM ÖZLEM ÇİNAR ÖZDEMİR, Assoc. Dr., Principal Investigator — Izmir Democracy University; CEMRE GÖRÜNMEZOĞLU, MSc, Principal Investigator — Izmir Democracy University; SADIK KIVANÇ METİN, Prof. Dr., Principal Investigator — Dokuz Eylul University; ECEM ÖZDEMİR, Principal Investigator — Dokuz Eylul University; EMEK NAZIM EKER, Principal Investigator — Dokuz Eylul University; ANIL GİRGİN, Principal Investigator — Dokuz Eylul University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kunimoto B, Cooling M, Gulliver W, Houghton P, Orsted H, Sibbald RG. Best practices for the prevention and treatment of venous leg ulcers. Ostomy Wound Manage. 2001 Feb;47(2):34-46, 48-50. PMID 11235498
- [Background] de Moura RM, Gomes Hde A, da Silva SL, Britto RR, Dias RC. Analysis of the physical and functional parameters of older adults with chronic venous disease. Arch Gerontol Geriatr. 2012 Nov-Dec;55(3):696-701. doi: 10.1016/j.archger.2012.05.005. Epub 2012 Jun 7. PMID 22682424
- [Background] Aydin G, Yeldan I, Akgul A, Ipek G. Effects of inspiratory muscle training versus calf muscle training on quality of life, pain, venous function and activity in patients with chronic venous insufficiency. J Vasc Surg Venous Lymphat Disord. 2022 Sep;10(5):1137-1146. doi: 10.1016/j.jvsv.2022.04.012. Epub 2022 Jun 14. PMID 35710091